CLINICAL TRIAL: NCT02718625
Title: A Randomized Controlled Trial of Enzymatic Debridement of Pressure Ulcers With Clostridial Collagenase Ointment (SANTYL®) or Hydrogel (SoloSite®)
Brief Title: Study of SANTYL® vs Hydrogel (SoloSite®) for Pressure Ulcers
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Business Decision
Sponsor: Smith & Nephew, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 017-101-09-036
Record Dates: First submitted 2016-03-18; First posted 2016-03-24 (Estimated); Results first posted 2020-03-10 (Actual); Last update posted 2020-03-10 (Actual); Status verified 2020-02

CONDITIONS: Pressure Ulcer
Keywords: Pressure Ulcers; Bed sores; Long-term care; Nursing home
MeSH Terms: conditions — Pressure Ulcer | interventions — Collagenases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Santyl (Experimental): Santyl collagenase ointment applied topically once per day for up to six weeks
  Interventions: Biological: Santyl
- SoloSite® (Active Comparator): SOLOSITE is a hydrogel wound dressing with preservatives. It can donate moisture to rehydrate non-viable tissue. It absorbs exudate while retaining its structure in the wound.
  Interventions: Biological: SoloSite®

INTERVENTIONS:
Biological: Santyl — Collagenase ointment applied topically
  Arms: Santyl
Biological: SoloSite® — SOLOSITE is a hydrogel wound dressing with preservatives. It can donate moisture to rehydrate non-viable tissue. It absorbs exudate while retaining its structure in the wound.
  Arms: SoloSite®

SUMMARY:
This study is designed to compare SANTYL® versus hydrogel (SoloSite®) in the treatment of pressure ulcers for participants in a long-term care facility. After meeting study criteria, participants will be randomly assigned for application of SANTYL® or SoloSite® to their pressure ulcer for up to 6 weeks. A study previously conducted showed that in the long-term care setting, the removal of dead skin (debridement) with SANTYL® resulted in more participants achieving complete debridement, more rapidly than when SoloSite® is used. The goal of the present study is to confirm the results of the earlier study, demonstrating superior debridement outcomes for pressure ulcers of patients in long-term care as compared to ulcers managed with SoloSite®.

ELIGIBILITY:
Inclusion Criteria -

1. Provide written informed consent, which will consist of reading, signing, and dating the informed consent document after the Investigator, sub-Investigator or other designated study staff member has explained the study procedures, risks, and contact information.
2. Eighteen (18) years of age or older, of either sex, and of any race.
3. Willing to comply with protocol instructions, including allowing all study assessments.
4. Subject is in-patient in a long-term care facility.
5. A pressure ulcer present with a surface area ≥ 1.0 cm2 and ≤ 64.0 cm2 confirmed using the ImageIQ EDCIQ mobile imaging system. Only one qualifying ulcer per subject will be selected for the study (selection based on greatest clinical need, as assessed by the Investigator).
6. The target ulcer must present with ≥85% necrotic, nonviable tissue as assessed by two independent image reviewers.
7. The target ulcer has not been previously treated with hydrogel (SoloSite®) or with SANTYL®. Prior ulcers at or near the same location may have been treated with these products.
8. No current infections requiring treatment with antibiotics (antibiotic use is permitted for the purpose of urinary tract infection prophylaxis, but this must be explicitly stated in the subject's chart).
9. Acceptable state of health and nutrition with pre-albumin levels of ≥ 10 mg/dL (0.10 g/L), per the Screening local lab report. This is not required if a pre-albumin test within range has been conducted within the last 30 days.
10. A hemoglobin A1c < 7.9% per the Screening local lab report. This is not required if a hemoglobin A1c test within range has been conducted within the last 30 days.
11. Have adequate pressure redistribution to the affected area or off-loading if the ulcer is on a lower extremity.
12. No known allergies or sensitivities to either test article or the dressings.

Women of child-bearing potential (those who are not premenarchal, not surgically sterilized [hysterectomy or bilateral oophorectomy], or not post-menopausal), may participate in the study if they meet the following condition:

-A negative urine pregnancy test at screening

Exclusion Criteria -

1. Undergoing therapy with another investigational agent within thirty (30) days of Study Visit 1, or planned participation overlapping with this study.
2. Current oral steroid treatment with a daily dose exceeding 5 mg.
3. Inability to comply with off-loading.
4. If the ulcer is on a lower extremity, inadequate arterial blood flow to the affected limb as evidenced by an ankle brachial index (ABI) <0.85.
5. Presence of callus requiring surgical debridement within 3 days of Study Visit 1.
6. Target ulcer with exposure of tendon, muscle or bone.
7. Medical condition that, in the opinion of the Investigator, would preclude safe subject participation in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2016-08 (Actual); Primary Completion 2017-03-09 (Actual); Study Completion 2017-03-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Herbert B Slade, MD, Study Chair — Smith & Nephew, Inc.; Jaime E Dickerson, PhD, Study Director — Smith & Nephew, Inc.; Martha Kelso, RN, Principal Investigator — Wound Care Plus
Locations (1):
- Lee's Summit, Missouri, United States

IPD SHARING:
Plan to Share IPD: Undecided

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study was conducted from 10October2016 to 09March2017. The study was cancelled by the sponsor due to low enrollment despite several attempts and measures to improve recruitment. Therefore, the study was not feasible to continue and an early termination was needed.
Period: Overall Study
Arm/Group | Santyl | SoloSite®
Started | 1 | 2
Completed | 1 | 0
Not Completed | 0 | 2
Not completed — Adverse Event | 0 | 1
Not completed — Termination of Study by Sponsor | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Santyl | SoloSite® | Total
Number analyzed (Participants) | 1 | 2 | 3
Age, Customized [Number; unit: years] — Population: Due to early study termination by Sponsor, data are presented by subject.
  years
    Subject 01-001: number analyzed (Participants) | 1 | 0 | 1
    Subject 01-001 | 74 |  | 74
    Subject 01-002: number analyzed (Participants) | 0 | 1 | 1
    Subject 01-002 |  | 58 | 58
    Subject 01-008: number analyzed (Participants) | 0 | 1 | 1
    Subject 01-008 |  | 46 | 46
Sex/Gender, Customized [Count of Participants; unit: Participants] — Population: Due to early study termination by Sponsor, data are presented by subject.
  Participants
    Subject 01-001: number analyzed (Participants) | 1 | 0 | 1
    Subject 01-001: Male | 0 |  | 0
    Subject 01-001: Female | 1 |  | 1
    Subject 01-002: number analyzed (Participants) | 0 | 1 | 1
    Subject 01-002: Male |  | 1 | 1
    Subject 01-002: Female |  | 0 | 0
    Subject 01-008: number analyzed (Participants) | 0 | 1 | 1
    Subject 01-008: Male |  | 1 | 1
    Subject 01-008: Female |  | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants] — Population: Due to early study termination by Sponsor, data are presented by subject.
  Participants
    Subject 01-001: number analyzed (Participants) | 1 | 0 | 1
    Subject 01-001: Hispanic or Latino | 0 |  | 0
    Subject 01-001: Not Hispanic or Latino | 1 |  | 1
    Subject 01-001: Unknown or Not Reported | 0 |  | 0
    Subject 01-002: number analyzed (Participants) | 0 | 1 | 1
    Subject 01-002: Hispanic or Latino |  | 0 | 0
    Subject 01-002: Not Hispanic or Latino |  | 1 | 1
    Subject 01-002: Unknown or Not Reported |  | 0 | 0
    Subject 01-008: number analyzed (Participants) | 0 | 1 | 1
    Subject 01-008: Hispanic or Latino |  | 0 | 0
    Subject 01-008: Not Hispanic or Latino |  | 1 | 1
    Subject 01-008: Unknown or Not Reported |  | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants] — Population: Due to early study termination by Sponsor, data are presented by subject.
  Participants
    Subject 01-001: number analyzed (Participants) | 1 | 0 | 1
    Subject 01-001: American Indian or Alaska Native | 0 |  | 0
    Subject 01-001: Asian | 0 |  | 0
    Subject 01-001: Native Hawaiian or Other Pacific Islander | 0 |  | 0
    Subject 01-001: Black or African American | 0 |  | 0
    Subject 01-001: White | 1 |  | 1
    Subject 01-001: More than one race | 0 |  | 0
    Subject 01-001: Unknown or Not Reported | 0 |  | 0
    Subject 01-002: number analyzed (Participants) | 0 | 1 | 1
    Subject 01-002: American Indian or Alaska Native |  | 0 | 0
    Subject 01-002: Asian |  | 0 | 0
    Subject 01-002: Native Hawaiian or Other Pacific Islander |  | 0 | 0
    Subject 01-002: Black or African American |  | 1 | 1
    Subject 01-002: White |  | 0 | 0
    Subject 01-002: More than one race |  | 0 | 0
    Subject 01-002: Unknown or Not Reported |  | 0 | 0
    Subject 01-008: number analyzed (Participants) | 0 | 1 | 1
    Subject 01-008: American Indian or Alaska Native |  | 0 | 0
    Subject 01-008: Asian |  | 0 | 0
    Subject 01-008: Native Hawaiian or Other Pacific Islander |  | 0 | 0
    Subject 01-008: Black or African American |  | 0 | 0
    Subject 01-008: White |  | 1 | 1
    Subject 01-008: More than one race |  | 0 | 0
    Subject 01-008: Unknown or Not Reported |  | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 1 | 2 | 3
Pressure Ulcer Scale for Healing (PUSH) Score [Number; unit: score on a scale] — Changes in wound status were to be measured by using the Pressure Ulcer Scale for Healing (PUSH) Tool. For baseline assessments at Visit 1, the target ulcer was to be scored based on length/width (from 0 cm^2 to >24 cm^2 on a scale of 1 to 10), exudate amount (from 'none' to 'heavy' on a scale of 0 to 3) , and tissue type ('closed' to 'necrotic tissue' on a scale of 0 to 4); from which a total PUSH score from the sum of scores for the three categories could be derived (ranging from 0 to 17). Higher scores indicated a worse response. Population: Due to early termination by Sponsor, no collective analyses were completed and data are presented by individual subject.
  score on a scale
    Subject 01-001 Visit 1 (V1) PUSH Length/Width: number analyzed (Participants) | 1 | 0 | 1
    Subject 01-001 Visit 1 (V1) PUSH Length/Width | NA — Due to early study termination by Sponsor, ulcer area measurements and scoring by independent reviewers did not occur; no PUSH length/width score was determined. |  | NA — Due to early study termination by Sponsor, ulcer area measurements and scoring by independent reviewers did not occur; no PUSH length/width score was determined.
    Subject 01-001 V1 PUSH Exudate Amount: number analyzed (Participants) | 1 | 0 | 1
    Subject 01-001 V1 PUSH Exudate Amount | 0 |  | 0
    Subject 01-001 V1 PUSH Tissue Type: number analyzed (Participants) | 1 | 0 | 1
    Subject 01-001 V1 PUSH Tissue Type | 4 |  | 4
    Subject 01-002 V1 PUSH Length/Width: number analyzed (Participants) | 0 | 1 | 1
    Subject 01-002 V1 PUSH Length/Width |  | NA — Due to early study termination by Sponsor, ulcer area measurements and scoring by independent reviewers did not occur; no PUSH length/width score was determined. | NA — Due to early study termination by Sponsor, ulcer area measurements and scoring by independent reviewers did not occur; no PUSH length/width score was determined.
    Subject 01-002 V1 PUSH Exudate Amount: number analyzed (Participants) | 0 | 1 | 1
    Subject 01-002 V1 PUSH Exudate Amount |  | 0 | 0
    Subject 01-002 V1 PUSH Tissue Type: number analyzed (Participants) | 0 | 1 | 1
    Subject 01-002 V1 PUSH Tissue Type |  | 4 | 4
    Subject 01-008 V1 PUSH Length/Width: number analyzed (Participants) | 0 | 1 | 1
    Subject 01-008 V1 PUSH Length/Width |  | NA — Due to early study termination by Sponsor, ulcer area measurements and scoring by independent reviewers did not occur; no PUSH length/width score was determined. | NA — Due to early study termination by Sponsor, ulcer area measurements and scoring by independent reviewers did not occur; no PUSH length/width score was determined.
    Subject 01-008 V1 PUSH Exudate Amount: number analyzed (Participants) | 0 | 1 | 1
    Subject 01-008 V1 PUSH Exudate Amount |  | 1 | 1
    Subject 01-008 V1 PUSH Tissue Type: number analyzed (Participants) | 0 | 1 | 1
    Subject 01-008 V1 PUSH Tissue Type |  | 3 | 3
Wound Bed Sore (WBS) Score [Number; unit: score on a scale] — Changes in wound status were to be measured by using the Wound Bed Sore (WBS) score. For the baseline assessment at Visit 1, 8 individual wound bed sore characteristics were scored, each on a scale of 0 to 2 (higher scores represented better outcomes), and then summed to derive the total WBS score (ranging from 0 to 16). Population: Due to early termination by Sponsor, no collective analyses were completed and data are presented by individual subject.
  score on a scale
    Subject 01-001 Visit 1 (V1) WBS Healing Edges: number analyzed (Participants) | 1 | 0 | 1
    Subject 01-001 Visit 1 (V1) WBS Healing Edges | 2 |  | 2
    Subject 01-001 V1 WBS Black Eschar: number analyzed (Participants) | 1 | 0 | 1
    Subject 01-001 V1 WBS Black Eschar | 0 |  | 0
    Subject 01-001 V1 WBS Greatest Wound Depth/Granul.: number analyzed (Participants) | 1 | 0 | 1
    Subject 01-001 V1 WBS Greatest Wound Depth/Granul. | 2 |  | 2
    Subject 01-001 V1 WBS Exudate Amount: number analyzed (Participants) | 1 | 0 | 1
    Subject 01-001 V1 WBS Exudate Amount | 2 |  | 2
    Subject 01-001 V1 WBS Edema: number analyzed (Participants) | 1 | 0 | 1
    Subject 01-001 V1 WBS Edema | 2 |  | 2
    Subject 01-001 V1 WBS Peri-Ulcer Dermatitis: number analyzed (Participants) | 1 | 0 | 1
    Subject 01-001 V1 WBS Peri-Ulcer Dermatitis | 2 |  | 2
    Subject 01-001 V1 WBS Peri-Ulcer Callus/Fibrosis: number analyzed (Participants) | 1 | 0 | 1
    Subject 01-001 V1 WBS Peri-Ulcer Callus/Fibrosis | 2 |  | 2
    Subject 01-001 V1 WBS Pink Ulcer Bed: number analyzed (Participants) | 1 | 0 | 1
    Subject 01-001 V1 WBS Pink Ulcer Bed | 2 |  | 2
    Subject 01-002 V1 WBS Healing Edges: number analyzed (Participants) | 0 | 1 | 1
    Subject 01-002 V1 WBS Healing Edges |  | 2 | 2
    Subject 01-002 V1 WBS Black Eschar: number analyzed (Participants) | 0 | 1 | 1
    Subject 01-002 V1 WBS Black Eschar |  | 0 | 0
    Subject 01-002 V1 WBS Greatest Wound Depth/Granul.: number analyzed (Participants) | 0 | 1 | 1
    Subject 01-002 V1 WBS Greatest Wound Depth/Granul. |  | 2 | 2
    Subject 01-002 V1 WBS Exudate Amount: number analyzed (Participants) | 0 | 1 | 1
    Subject 01-002 V1 WBS Exudate Amount |  | 2 | 2
    Subject 01-002 V1 WBS Edema: number analyzed (Participants) | 0 | 1 | 1
    Subject 01-002 V1 WBS Edema |  | 2 | 2
    Subject 01-002 V1 WBS Peri-Ulcer Dermatitis: number analyzed (Participants) | 0 | 1 | 1
    Subject 01-002 V1 WBS Peri-Ulcer Dermatitis |  | 2 | 2
    Subject 01-002 V1 WBS Peri-Ulcer Callus/Fibrosis: number analyzed (Participants) | 0 | 1 | 1
    Subject 01-002 V1 WBS Peri-Ulcer Callus/Fibrosis |  | 2 | 2
    Subject 01-002 V1 WBS Pink Ulcer Bed: number analyzed (Participants) | 0 | 1 | 1
    Subject 01-002 V1 WBS Pink Ulcer Bed |  | 2 | 2
    Subject 01-008 V1 WBS Healing Edges: number analyzed (Participants) | 0 | 1 | 1
    Subject 01-008 V1 WBS Healing Edges |  | 1 | 1
    Subject 01-008 V1 WBS Black Eschar: number analyzed (Participants) | 0 | 1 | 1
    Subject 01-008 V1 WBS Black Eschar |  | 2 | 2
    Subject 01-008 V1 WBS Greatest Wound Depth/Granul.: number analyzed (Participants) | 0 | 1 | 1
    Subject 01-008 V1 WBS Greatest Wound Depth/Granul. |  | 0 | 0
    Subject 01-008 V1 WBS Exudate Amount: number analyzed (Participants) | 0 | 1 | 1
    Subject 01-008 V1 WBS Exudate Amount |  | 2 | 2
    Subject 01-008 V1 WBS Edema: number analyzed (Participants) | 0 | 1 | 1
    Subject 01-008 V1 WBS Edema |  | 2 | 2
    Subject 01-008 V1 WBS Peri-Ulcer Dermatitis: number analyzed (Participants) | 0 | 1 | 1
    Subject 01-008 V1 WBS Peri-Ulcer Dermatitis |  | 2 | 2
    Subject 01-008 V1 WBS Peri-Ulcer Callus/Fibrosis: number analyzed (Participants) | 0 | 1 | 1
    Subject 01-008 V1 WBS Peri-Ulcer Callus/Fibrosis |  | 2 | 2
    Subject 01-008 V1 WBS Pink Ulcer Bed: number analyzed (Participants) | 0 | 1 | 1
    Subject 01-008 V1 WBS Pink Ulcer Bed |  | 2 | 2

OUTCOME MEASURES:

1. Primary Outcome: Proportion of Ulcers With Complete Debridement
Description: For purposes of the primary analysis, the status of complete debridement was to be assessed from photographs by two independent reviewers.
Time Frame: 6 weeks
Population: Due to early study termination by Sponsor, complete debridement assessment by independent review of ulcer photographs did not take place.
Arm/Group | Santyl | SoloSite®
Number analyzed (Participants) | 0 | 0

2. Secondary Outcome: Time in Days to Complete Debridement
Description: For purposes of this secondary analysis, the time (in days) to achieve complete debridement (as defined in the primary analysis) was to be calculated from the date of randomization visit to the date of which the subject's ulcer was deemed to have achieved complete debridement.
Time Frame: 6 weeks
Population: Due to early study termination by Sponsor, complete debridement assessment by independent review of ulcer photographs did not take place and time (in days) to complete debridement was not calculated.
Arm/Group | Santyl | SoloSite®
Number analyzed (Participants) | 0 | 0

3. Secondary Outcome: Percentage Reduction in Non-viable Tissue
Description: For purposes of this secondary analysis, the assessment of percentage of non-viable necrotic tissue was to be assessed based on photograph review by two independent reviewers, with the reduction calculated as: percentage of non-viable necrotic tissue at Visit 1 - percentage of non-viable necrotic tissue at Visit 7.
Time Frame: 6 weeks
Population: Due to early study termination by Sponsor, the assessment of ulcer photographs by two independent reviewers did not take place; thus, the analysis of this secondary outcome was not possible.
Arm/Group | Santyl | SoloSite®
Number analyzed (Participants) | 0 | 0

4. Secondary Outcome: Percentage Reduction in Ulcer Area
Description: For purposes of this secondary analysis, the percentage reduction in ulcer area was to be measured during ulcer photograph review by two independent reviewers, using the ImageIQ EDCIQ mobile imaging system, with the reduction calculated as: ([ulcer area at Visit 1 - ulcer area at Visit 7 / ulcer area at Visit 1] x 100).
Time Frame: 6 weeks
Population: Due to early study termination by Sponsor, the independent reviewers' assessment of ulcer photographs did not take place; thus, the analysis of this secondary outcome was not possible.
Arm/Group | Santyl | SoloSite®
Number analyzed (Participants) | 0 | 0

5. Secondary Outcome: Pressure Ulcer Scale for Healing (PUSH) Score
Description: For purposes of this secondary analysis, changes in wound status were to be measured by using the Pressure Ulcer Scale for Healing (PUSH) Tool. At Visits 1 and 7, the target ulcer was to be scored based on length/width (from 0 cm^2 to >24 cm^2 on a scale of 1 to 10), exudate amount (from 'none' to 'heavy' on a scale of 0 to 3) , and tissue type ('closed' to 'necrotic tissue' on a scale of 0 to 4); from which a total PUSH score from the sum of scores for the three categories could be derived (ranging from 0 to 17). Higher scores indicated a worse response. The reduction in PUSH individual sub-scores and total PUSH scores were calculated as: (PUSH Score at Visit 1 - Push Score at Visit 7/Exit).
Time Frame: 6 weeks
Population: Due to early study termination by Sponsor, only one subject completed the study and underwent Visit 7/Exit assessments (in the Santyl group). Ulcer area measurements and scoring by independent reviewers did not occur; no PUSH length/width score was determined. No analyses were done and individual data are presented for the single completed subject.
Measure: Number; unit: score on a scale
Arm/Group | Santyl | SoloSite®
Number analyzed (Participants) | 1 | 0
score on a scale
  Subject 01-001 Visit 7/Exit (V7) PUSH Length/Width: number analyzed (Participants) | 0 | 0
  Subject 01-001 V7 PUSH Exudate Amount | 1 |
  Subject 01-001 V7 PUSH Tissue Type | 4 |

6. Secondary Outcome: Wound Bed Sore (WBS) Score
Description: For purposes of this secondary analysis, changes in wound status were to be measured by using the Wound Bed Sore (WBS) score. At Visits 1 and 7, eight individual wound bed sore characteristics were scored, each on a scale of 0 to 2 (higher scores represented better outcomes), and then summed to derive the total WBS score (ranging from 0 to 16). The reduction in total WBS scores were calculated as: (Total WBS Score at Visit 1 - Total WBS Score at Visit 7/Exit).
Time Frame: 6 weeks
Population: Due to early study termination by Sponsor, only one subject completed the study and underwent Visit 7/Exit assessments (in the Santyl group). No analyses were done and individual data are presented for the single completed subject.
Measure: Number; unit: score on a scale
Arm/Group | Santyl | SoloSite®
Number analyzed (Participants) | 1 | 0
score on a scale
  Subject 01-001 Visit 7/Exit (V7) WBS Healing Edges | 2 |
  Subject 01-001 V7 WBS Black Eschar | 0 |
  Subject 01-001 V7 WBS Greatest Wound Depth/Granul. | 1 |
  Subject 01-001 V7 WBS Exudate Amount | 2 |
  Subject 01-001 V7 WBS Edema | 2 |
  Subject 01-001 V7 WBS Peri-Ulcer Dermatitis | 2 |
  Subject 01-001 V7 WBS Peri-Ulcer Callus/Fibrosis | 2 |
  Subject 01-001 V7 WBS Pink Ulcer Bed | 0 |

ADVERSE EVENTS:
Time Frame: Approximately 7 weeks (i.e., study participation duration)
Arm/Group | Santyl | SoloSite®
All-Cause Mortality (participants affected / at risk) | 0/1 | 0/2
Serious Adverse Events (participants affected / at risk) | 0/1 | 1/2
Other Adverse Events (participants affected / at risk) | 0/1 | 0/2
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Santyl (N=1) | SoloSite® (N=2)
Altered Mental Status (General disorders) | 0 (0) | 1 (1) — Patient was experiencing altered mental status and was found to have a decreased level of consciousness by facility staff. Facility staff reported that the patient was unable to answer questions appropriately and was not speaking coherently.

LIMITATIONS AND CAVEATS:
Due to the early termination of the study by the sponsor and the number of subjects enrolled, data were not analyzed or summarized and were only listed by subject. The safety and efficacy of Santyl could not be assessed based on this study.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-05-05): https://cdn.clinicaltrials.gov/large-docs/25/NCT02718625/Prot_SAP_000.pdf